CLINICAL TRIAL: NCT04551937
Title: The Effects of Prebiotics on Behavioral and Biological Markers of Cognition and Stress
Brief Title: Effects of Prebiotics on Cognition and Health
Acronym: EPOCH-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Hannah Holscher, Assistant Professor of Nutrition, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 16840
Record Dates: First submitted 2018-07-06; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Physiological Stress; Cognitive Change; Gastrointestinal Health
MeSH Terms: interventions — Milk; Prebiotics

STUDY DESIGN:
Intervention Model Description: Participants will pass through 2 arms, control and prebiotic, in a randomized, counterbalanced order.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind (participant and investigative team)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): 4-5 week period where participant will consume control beverage
  Interventions: Other: Lactose Free 1% Milk
- Prebiotic (Experimental): 4-5 week period where participant will consume the intervention beverage
  Interventions: Other: Lactose Free 1% Milk + 10 g prebiotic

INTERVENTIONS:
Other: Lactose Free 1% Milk — 8 oz of study beverage daily
  Other Names: Control
  Arms: Control
Other: Lactose Free 1% Milk + 10 g prebiotic — 8 oz of study beverage supplemented with 5 grams of fructooligosaccharide and 5 grams of galactooligosaccharide
  Arms: Prebiotic

SUMMARY:
This research intervention aims to examine the effects of prebiotic consumption on changes in behavioral and biological measures of cognition and stress among adults.

DETAILED DESCRIPTION:
Evidence-based dietary strategies provide behavioral means benefiting physical and cognitive function. Pertinent to the proposed work, dietary intake has been recently shown to have the potential to directly influence the gut microbiota composition as well as brain function. Specifically, the consumption of prebiotics or fibers metabolized by gut bacteria may also play a role. These foods are readily available in the marketplace, however, their implications for physical and cognitive function are not clear. Accordingly, the proposed study aims to investigate effects of prebiotic beverage consumption on changes in behavioral and biological measures of cognition and stress among adults.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Between the ages of 25-45 years at the time of consent
* BMI ≥18.5 kg/m2
* Normal or corrected-to-normal vision based on the minimal 20/20 standard in order to complete the cognitive task.
* Ability to drop-off fecal sample within 15 minutes of defecation

Exclusion Criteria:

* Current pregnancy or lactation
* Tobacco use
* Dairy allergy or intolerance
* Prior diagnosis of metabolic and gastrointestinal disease (cardiovascular disease and type 1 or type 2 diabetes, chronic constipation, diarrhea, Crohn's disease, celiac disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, hepatitis, HIV, cancer, etc.)
* Prior diagnosis of cognitive or physical disability, including ADHD, severe asthma, epilepsy, chronic kidney disease
* Use of any anti-psychotic, anti-depressant, antianxiety, or ADD/ADHD medications
* Use of medications that alter normal bowel function and metabolism (e.g., recent antibiotic use, laxatives, enemas, anti-diarrheal agents, narcotics, antispasmodics, diuretics, anticonvulsants).
* Prior malabsorptive bariatric surgery (i.e. gastric bypass, sleeve gastrectomy) or restrictive bariatric surgery (i.e. adjustable gastric band)

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Biological markers of stress | 4-5 weeks
  Changes in 24-hour urinary cortisol, inflammatory markers (e.g. IL-6, CRP).
Behavioral markers of stress | 4-5 weeks
  Change in reported questionnaire responses specific to depression, stress, and anxiety using the Depression, Anxiety, and Stress (DASS) Questionnaire.

SECONDARY OUTCOMES:
Gastrointestinal Microbiota composition | 4-5 weeks
  Impact on bacterial genera abundances.
Gastrointestinal microbiota beta-diversity | 4-5 weeks
  Impact on beta-diversity measures
Gastrointestinal Microbiota alpha-diversity | 4-5 weeks
  Impact on alpha-diversity measures
Cognitive function | 4-5 weeks
  Computer tasks will be used to assess working memory, interference control, cognitive flexibility, and hippocampal function/relational memory
Sleep | 4-5 weeks
  The Pittsburg Sleep Quality Index (PSQI) will also be used to assess sleep, as will actigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Holscher, PhD, RD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mysonhimer AR, Cannavale CN, Bailey MA, Khan NA, Holscher HD. Prebiotic Consumption Alters Microbiota but Not Biological Markers of Stress and Inflammation or Mental Health Symptoms in Healthy Adults: A Randomized, Controlled, Crossover Trial. J Nutr. 2023 Apr;153(4):1283-1296. doi: 10.1016/j.tjnut.2023.02.015. Epub 2023 Feb 24. PMID 36841506